CLINICAL TRIAL: NCT04632056
Title: A 52-weeks Observational Study to Evaluate the Safety of Brolucizumab (6mg) in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: A 52-weeks Observational Study to Evaluate the Safety of Brolucizumab in Patients With nAMD
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258A1401
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Japan; brolucizumab; neovascular age-related macular degeneration; (nAMD); non-interventional study; post-marketing surveillance
MeSH Terms: interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Beovu: Brolucizumab (Genetical Recombination) 6 mg (0.05 mL) was administered by intravitreal injection every 4 weeks for the first three doses(loading phase). In the following maintenance phase, Brolucizumab was basically administered every 12 weeks. The interval between treatments was adjusted as appropriate according to the symptoms. The interval between two doses was not to be shorter than 8 weeks
  Interventions: Drug: Beovu

INTERVENTIONS:
Drug: Beovu — There is no treatment allocation. Patients administered Beovu by prescription that have started before inclusion of the patient into the study were enrolled.
  Other Names: Brolucizumab

SUMMARY:
This study was a prospective, uncontrolled, central registration system, multicenter, domestic observational study (special drug-use surveillance) to evaluate the safety of 52-week clinical treatment with Beovu kit for intravitreal injection in nAMD patients.

DETAILED DESCRIPTION:
The observational period was 1 year (52 weeks) from the first brolucizumab administration in the primary treated eye.

However, if brolucizumab was discontinued in the primary treated eye and if the treatment was discontinued less than 52 weeks observation period, the observation period was to be up to 90 days after the last dose of this drug. This was set in order to collect data as much as possible based on the clinical effect of the drug. If 30 days after the last dose of this drug in a discontinued patient exceeds 52 weeks of the observation period, the patient was to be monitored for adverse events until 30 days after the last dose of this drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written consent to cooperate in this study before treatment with Beovu kit for intravitreal injection
2. Patients using Beovu kit for intravitreal injection for the first time for the following indication:

   * Indication: age-related macular degeneration with subfoveal choroidal neovascularization

Exclusion Criteria:

1. Patients with a history of treatment with a drug containing the same ingredient (brolucizumab; investigational drug or post-marketing clinical study drug) as Beovu kit for intravitreal injection

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population was patients using Beovu kit for intravitreal injection for nAMD with subfoveal CNV
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events in the eyes on therapy | 52 weeks
  Number of patients with adverse events (AEs) in the eyes on therapy were reported
Number of patients with adverse events in other parts of the body (non-ocular) | 52 weeks
  Number of patients with adverse events (AEs) in other parts of the body (non-ocular) were reported

SECONDARY OUTCOMES:
Number of patients with serious adverse events (SAEs) and adverse reactions (ADRs) in the eyes on therapy | 52 weeks
  A SAE is defined as an AE whose description suggests that it is serious or whose outcome is fatal.
  An adverse reaction is defined as an adverse event that is suspected by the investigator to be causally related to Beovu or administration procedures, or whose causality is not recorded.
Number of patients with SAEs and ADRs in other parts of the body (non-ocular) | 52 weeks
  A SAE is defined as an AE whose description suggests that it is serious or whose outcome is fatal.
  An adverse reaction is defined as an adverse event that is suspected by the investigator to be causally related to Beovu or administration procedures, or whose causality is not recorded.
Number of patients with adverse events, SAEs, ADRs and serious ADRs corresponding to the safety specifications | 52 weeks
  The following events were chosen as the safety specifications for this study that should be investigated:
  * Intraocular inflammation
  * Endophthalmitis
  * Increased intraocular pressure
  * Retinal pigment epithelial tear
  * Retinal detachment and retinal tear
  * Retinal artery embolic events
  * Non-ocular arterial thromboembolic events
  * Retinal vasculitis and retinal vascular occlusion
Incidence of adverse events by risk factor of the safety specifications (primary treated eyes only) | 52 weeks
  Incidence of adverse events by risk factor of the safety specifications (primary treated eyes only) were reported
Proportion of patients with visual acuity (VA) worsening | 52 weeks
  Visual acuity commonly refers to the clarity of vision
Data on Beovu administration in the induction phase and maintenance phase | 52 weeks
  For data on Beovu administration (dosing duration, dosing frequency) in the primary treated eye and the secondary primary eyes in the safety analysis set, summary statistics were calculated respectively. The same calculation applied to data on administration respectively for the induction period and the maintenance period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (56):
- Japan (56):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyohashi, Aichi-ken
  - Novartis Investigative Site, Urayasu, Chiba
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Hakodate, Hokkaido
  - Novartis Investigative Site, Hakodat, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kakogawa-shi, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Ishioka, Ibaraki
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Yokkaichi, Mie-ken
  - Novartis Investigative Site, Kesennuma, Miyagi
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Miyakonojō, Miyazaki
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Nakagami, Okinawa
  - Novartis Investigative Site, Urazoe, Okinawa
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Saitama-shi, Saitama
  - Novartis Investigative Site, Ohtsu-city, Shiga
  - Novartis Investigative Site, Oda, Shimane
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Izunokuni, Shizuoka
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Musashino, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Nagasaki
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258A1401 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18111